CLINICAL TRIAL: NCT00121160
Title: Can Stress Management Improve Vaccine Immune Response
Brief Title: Health SMART (Stress Management and Relaxation Training) to Improve Vaccine Immune Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Bonnie A. McGregor, PhD / Assistant Member, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-6003; NCI-K01-CA107085-01
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Psychological Stress
Keywords: immune response to vaccines; stress management; breast cancer
MeSH Terms: conditions — Stress, Psychological; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management (CBSM) group intervention — Participants will meet in closed, structured groups of 4 to 6 women for ten weekly, 2-hour group sessions. The intervention employs CBSM techniques interwoven with information in a supportive group format. The information portion of the intervention focuses on learning to cope with daily stressors, and learning about optimal use of social support. Group members and group leaders are used as role models for effective coping and the use of social support. The groups also encourage emotional expression and provide an opportunity to practice techniques learned in the group and experience social support. Avoidance coping is discouraged, and acceptance and reframing are instead encouraged as coping responses. Health behavior change, framed as a coping technique, will also be discussed using motivational interviewing techniques. Each week participants also experience a different relaxation technique. The goal of the CBSM intervention is thus to reduce distress through a variety of techniques.

SUMMARY:
The proposed investigation will conduct a randomized, clinical trial to test the efficacy of a cognitive behavioral stress management (CBSM) group intervention on immune response to vaccine and distress among women at elevated risk for breast cancer.

Hypothesis 1: Women who participate in the CBSM intervention will have a larger primary and secondary antibody response to vaccines compared to women in the comparison group.

Hypothesis 2: Women who participate in a 10-week CBSM group intervention will report lower levels of distress immediately after and 6 months after the intervention compared to women in the comparison group.

DETAILED DESCRIPTION:
Chronic stress can impair immune function, including immune response to vaccines. This has important implications for cancer control and prevention because tumor vaccines are emerging as tools for cancer treatment and prevention, and the cohort that would benefit from the vaccines is likely to be stressed. Women at elevated risk for breast cancer experience significant levels of distress that have been associated with immune function decrements. Interventions to treat distress-related immune decrements among these women are needed because these women will be among the first candidates for breast cancer vaccines. In theory, stress-management interventions should improve immune function and response to vaccines, but the findings to date are mixed, in part because most intervention studies have been done with medical patients who by nature have immune confounds. Thus, it is unknown how stress management interventions affect immune function in stressed but otherwise healthy people, such as women at elevated risk for breast cancer.

Comparison: Women will be randomly assigned to a 10-week structured, CBSM intervention or a wait-list comparison group with delay participation in the intervention. The comparison group will be offered the full CBSM intervention after all assessment time points have been completed.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-60 years
* Family history of breast cancer
* Fluent in English
* Working phone
* Working address
* Plan to live in the area for one year

Exclusion Criteria:

* Prior cancer diagnosis (except non-melanoma skin cancer)
* Current major depressive episode
* History of Bipolar Disorder or Schizophrenia
* History of autoimmune disease
* History of Hepatitis A or HA vaccination
* Current infectious disease
* Use of immune modulating drugs

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Independent sample t-test will be used to compare 1) antibody change scores from before to after the first and second dose of vaccine, and 2) distress change scores from before to after the intervention | length of protocol

SECONDARY OUTCOMES:
Multiple regression analyzes will be used to test changes in cortisol and changes in perceived risk of breast cancer; coping or social support mediate the effects of the intervention on antibody response to vaccine and distress | length of protocol

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie A. McGregor, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] McEwen BS. Protective and damaging effects of stress mediators. N Engl J Med. 1998 Jan 15;338(3):171-9. doi: 10.1056/NEJM199801153380307. No abstract available. PMID 9428819
- [Background] Reichlin S. Alternative pathways of neural control of the immune process. Ann N Y Acad Sci. 1998 May 1;840:301-16. doi: 10.1111/j.1749-6632.1998.tb09570.x. PMID 9629258
- [Background] Cohen S, Miller GE, Rabin BS. Psychological stress and antibody response to immunization: a critical review of the human literature. Psychosom Med. 2001 Jan-Feb;63(1):7-18. doi: 10.1097/00006842-200101000-00002. PMID 11211068
- [Background] Miller GE, Cohen S. Psychological interventions and the immune system: a meta-analytic review and critique. Health Psychol. 2001 Jan;20(1):47-63. doi: 10.1037//0278-6133.20.1.47. PMID 11199066
- [Background] Cohen M, Klein E, Kuten A, Fried G, Zinder O, Pollack S. Increased emotional distress in daughters of breast cancer patients is associated with decreased natural cytotoxic activity, elevated levels of stress hormones and decreased secretion of Th1 cytokines. Int J Cancer. 2002 Jul 20;100(3):347-54. doi: 10.1002/ijc.10488. PMID 12115552
- [Background] Lerman C, Kash K, Stefanek M. Younger women at increased risk for breast cancer: perceived risk, psychological well-being, and surveillance behavior. J Natl Cancer Inst Monogr. 1994;(16):171-6. PMID 7999461
- [Background] Kash KM, Holland JC, Halper MS, Miller DG. Psychological distress and surveillance behaviors of women with a family history of breast cancer. J Natl Cancer Inst. 1992 Jan 1;84(1):24-30. doi: 10.1093/jnci/84.1.24. PMID 1738170
- [Background] Lloyd S, Watson M, Waites B, Meyer L, Eeles R, Ebbs S, Tylee A. Familial breast cancer: a controlled study of risk perception, psychological morbidity and health beliefs in women attending for genetic counselling. Br J Cancer. 1996 Aug;74(3):482-7. doi: 10.1038/bjc.1996.387. PMID 8695370
- [Background] Hopwood P, Keeling F, Long A, Pool C, Evans G, Howell A. Psychological support needs for women at high genetic risk of breast cancer: some preliminary indicators. Psychooncology. 1998 Sep-Oct;7(5):402-12. doi: 10.1002/(SICI)1099-1611(1998090)7:53.0.CO;2-X. PMID 9809331
- [Background] Erblich J, Bovbjerg DH, Valdimarsdottir HB. Looking forward and back: distress among women at familial risk for breast cancer. Ann Behav Med. 2000 Winter;22(1):53-9. doi: 10.1007/BF02895167. PMID 10892528
- [Background] Decruyenaere M, Evers-Kiebooms G, Welkenhuysen M, Denayer L, Claes E. Cognitive representations of breast cancer, emotional distress and preventive health behaviour: a theoretical perspective. Psychooncology. 2000 Nov-Dec;9(6):528-36. doi: 10.1002/1099-1611(200011/12)9:63.0.co;2-#. PMID 11180588
- [Derived] McGregor BA, Dolan ED, Murphy KM, Sannes TS, Highland KB, Albano DL, Ward AA, Charbonneau AM, Redman MW, Ceballos RM. Cognitive Behavioral Stress Management for Healthy Women at Risk for Breast Cancer: a Novel Application of a Proven Intervention. Ann Behav Med. 2015 Dec;49(6):873-84. doi: 10.1007/s12160-015-9726-z. PMID 26290001